CLINICAL TRIAL: NCT02030678
Title: To Evaluate the Clinical Effect of Irinotecan Monotherapy in Treatment of Local Recurrence or Metastatic Breast Cancer Patients Who Accepted at Least 2 Kinds of Chemotherapy Regimens Including Antharcycline or Taxanes.
Brief Title: A Phase II Study of Irinotecan in 3 Line or More Therapy in Local Recurrence or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Sun Tao, Director of Oncology, Liaoning Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STao
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Stage IIIB, IV, Recurrent, and Metastatic Breast Cancer
MeSH Terms: conditions — Recurrence; Breast Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- irinotecan Hydrochloride (Experimental): Irinotecan monotherapy (trade name: Aili; batches 180103AG [40 mg] and 171231AG [100 mg]) will be administered intravenously at a dose of 100 mg/m2 on days 1 and 8 of each 3-week cycle.
  Interventions: Drug: irinotecan

INTERVENTIONS:
Drug: irinotecan — Irinotecan monotherapy (trade name: Aili; batches 180103AG [40 mg] and 171231AG [100 mg]) will be administered intravenously at a dose of 100 mg/m2 on days 1 and 8 of each 3-week cycle.
  Other Names: Kaiputuo

SUMMARY:
A phase II study of irinotecan in 3 line or more therapy in local recurrence or metastatic breast cancer. Evaluate the effect and safety of irinotecan in local recurrence or Metastatic breast cancer patients who recieved anthracycline or taxane drugs. The primary endpoint is Disease Control Rate and Progression free survival. The second endpoint is 3 or 4 grade Adverse Events 、overall survival.All the patients will recieve this therapy till disease progress or other occurrence of withdrawal standards.

DETAILED DESCRIPTION:
A phase II study of irinotecan in 3 line or more therapy in local recurrence or metastatic breast cancer. Evaluate the effect and safety of irinotecan in local recurrence or Metastatic breast cancer patients who recieved anthracycline or taxane drugs. The primary endpoint is Disease Control Rate and Progression free survival. The second endpoint is 3 or 4 grade Adverse Events 、overall survival. irinotecan 100mg/m2,iv,day1,day8,every 3cycles.If no AE happens, increase irinotecan dose to125mg/m2 at the second cycle.All the patients will recieve this therapy till disease progress or other occurrence of withdrawal standards.

ELIGIBILITY:
Inclusion Criteria:

* Mestatic breast cancer patients whose disease recurrent after using anthracycline or taxane drugs

Exclusion Criteria:

* Heart Disease.etc

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate | 3cycles (21days/cycle)
  Disease Control Rate:Completely Response+Partial Response+Stable Disease

CONTACTS AND LOCATIONS:
Overall Officials: Tao Sun, Doctor, Principal Investigator — Liaoning Cancer Hospital & Institute
Locations (1):
- SunTao, Shenyang, Liaoning, China